CLINICAL TRIAL: NCT03066674
Title: Effect of the Hands- on McKenzie Program on Derangement Syndrome in Sub-acute and Chronic Low Back Pain
Brief Title: Effect of the Hands- on McKenzie Program on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Lina Abdullah AL-Banawi, Physical Therapist, Imam Abdulrahman Bin Faisal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-03-178
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie group (Experimental): This group will receive Hand-on technique on the lumbar spine.
  Interventions: Other: McKenzie group
- Control group (Experimental): The Group will not receive Hand-on technique on the lumbar spine.
  Interventions: Other: Control group

INTERVENTIONS:
Other: McKenzie group — Mobilization for lumbar spine,TENS,Exercises,Postural education ,Home exercises program.
  Arms: McKenzie group
Other: Control group — TENS,Exercises,Postural education ,Home exercises program.
  Other Names: without any Hand -on Technique.
  Arms: Control group

SUMMARY:
Low back pain (LBP) is one of most prevalent types of musculoskeletal pain and is strongly related to disability. The McKenzie method is one of most popular treatment options for LBP.

The objectives of this study are to determine the effect of the hands-on McKenzie program on pain, disability, spine mobility, and posture deviations in subjects with derangement low back pain.

DETAILED DESCRIPTION:
Thirty eight patients with sub-acute and chronic LBP will be randomly assigned to the McKenzie group (MG) or the control group (CG). The MG will perform exercises with the hands-on procedure (three sessions per week) for two weeks, while the CG will perform only exercises for two weeks. Both groups will do a home exercise program. The outcome assessments will measure pain by the Pain Numerical Rating Scale (NPRS), the level of disability through the Oswestry Disability Index (ODI), spine mobility by range of motion (ROM) for the lumbar spine, and the centralization of symptoms and the postural alternation by postural analysis grid (PAG). By using SPSS version 20, a paired t-test will be use to study the effect of the McKenzie program before and after treatment. An independent t-test will be used to study the significance between the two groups.

ELIGIBILITY:
Inclusion Criteria:

- The patients will be age from 18 to 60 years old, and have LBP with or without leg pain, lasting from seven weeks to 12 weeks or more. Additional criteria include recurrent LBP, demonstrating a DP during the mechanical assessment , The subjects have a BMI of normal (17 to 23.9) or overweight (24 to 28.9). Patient is Eligible.

Exclusion Criteria:

Participants who are underweight (BMI < 18.5) or obese (BMI ≥ 30) will be excluded . Those with contraindications to physical exercise according to the guidelines of the American College of Sports Medicine , such as those with serious spinal pathologies (fractures, tumours, and inflammatory diseases, such as ankylosing spondylitis), nerve root compromise (e.g., cauda equine syndrome), severe cardiopulmonary diseases,SCD, or pregnancy will be excluded.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale (PNRS). | Two weeks
  For assessing the pain in the low back.

SECONDARY OUTCOMES:
Spine mobility | Two weeks
  In the flexion/extension/rotation and side bending(Right -Left)
Centralization or non-centralizer (Peripheralization) of patient symptoms. | Two weeks.
  Using the body chart.
Postural alterations. | Two weeks
  It is measure by Postural Analysis Grid (PAG) and software
Disability associated with LBP | Two weeks
  It is measure by The Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: LINA A ALBANAWI, MASTER, Study Chair — Imam Abdulrahman Bin Faisal University

IPD SHARING:
Plan to Share IPD: Undecided